CLINICAL TRIAL: NCT00486954
Title: A Randomized, Multicenter, Open-label, Phase III Study of Lapatinib (GW572016) in Combination With Weekly Paclitaxel Versus Weekly Paclitaxel Alone in the Second Line Treatment of ErbB2 Amplified Advanced Gastric Cancer
Brief Title: Lapatinib in Combination With Weekly Paclitaxel in Patients With ErbB2 Amplified Advanced Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104578
Record Dates: First submitted 2007-06-13; First posted 2007-06-15 (Estimated); Results first posted 2013-02-07 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-01

CONDITIONS: Neoplasms, Gastrointestinal Tract
Keywords: lapatinib; paclitaxel; ErbB2; Gastric cancer; Advanced gastric cancer
MeSH Terms: conditions — Neoplasms; Stomach Neoplasms | interventions — Lapatinib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paclitaxel plus Lapatinib (Experimental): 6 pills of lapatinib at 250 mg each once daily and infusion of paclitaxel at 80 mglm2 weekly
  Interventions: Drug: Lapatinib; Drug: Paclitaxel
- Paclitaxel alone (Active Comparator): Infusion of paclitaxel at 80 mglm2 weekly
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Lapatinib — 6 pills at 250 mg each once daily
  Other Names: Lapatinib: Tykerb; Tyverb
  Arms: Paclitaxel plus Lapatinib
Drug: Paclitaxel — Infusion at 80 mg/m2 weekly

SUMMARY:
EGF104578 is two-part study (Pilot part/Randomized part).Pilot part is designed to find the optimal (best) doses of lapatinib and paclitaxel when given together,Randomized part is designed to evaluate the overall survival in patients receiving lapatinib and paclitaxel compared to patients receiving only paclitaxel.

ELIGIBILITY:
Inclusion criteria:

Specific Information regarding warnings, precautions, contraindications, adverse events, and other pertinent information on the investigational product that may impact subject eligibility is provided in the Investigator's Brochure (IB) Pilot Part

Subjects eligible for enrollment in the Pilot Part of the study must meet all of the following criteria:

* Signed informed consent
* Male or female; ≥ 20 years (at the time of giving consent)
* Any histologically or cytologically confirmed gastric carcinoma independent of tumor ErbB2 status
* Subjects who have received one prior regimen for gastric carcinoma and developed disease progression or recurrence. The regimen must have contained 5-fluoropyrimidine and/or cisplatin
* Left ventricular ejection fraction (LVEF) within institutional range of normal as measured by echocardiogram (ECHO). Multigated acquisition (MUGA) scans will be accepted in cases where an echocardiogram cannot be performed or is inconclusive (LVEF of ≥50% required if normal range of LVEF is not provided by institution)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1
* Able to swallow and retain oral medication
* Women and men with potential to have children must be willing to practice acceptable methods of birth control during the study
* Washout period from the prior last therapy as follows; Chemotherapy (except for agents below) 4 weeks (I.V) Chemotherapy (except for agents below) 2 weeks (P.O) Trastuzumab, Bevacizumab 4 weeks Mitomycin-C, nitrosourea 6 weeks Radiotherapy, Immunotherapy, Biologic therapy and Surgery (except for minor surgical procedure) 2 weeks
* Willing to complete all screening assessments as outlined in the protocol
* Adequate organ function as defined in Table 2 Baseline Laboratory Values
* Able to be hospitalized for PK analysis during cycle 1
* Life expectancy of at least 12 weeks from the first dose of study treatment)

Randomized Part

Subjects eligible for enrollment in the Randomized Part of the study must meet all of the following criteria:

* Signed informed consent
* Male or female; ≥ 20 years (at the time of giving consent)
* Histologically or cytologically confirmed gastric carcinoma with documented amplification of ErbB2 by fluorescence in situ hybridization (FISH) in primary or metastatic tumor tissue
* Subjects who received one prior regimen for gastric carcinoma and defined as progression disease. The regimen must be containing 5-fluoropyrimidine and/or cisplatin
* Measurable lesion(s) according to RECIST (Response Evaluation Criteria in Solid Tumors)
* Left ventricular ejection fraction (LVEF) within institutional range of normal as measured by echocardiogram. MUGA scans will be accepted in cases where an echocardiogram cannot be performed or is inconclusive (LVEF of ≥50% required if normal range of LVEF is not provided by institution)
* ECOG Performance Status of 0 to 1
* Able to swallow and retain oral medication
* Archived (or Biopsy ) tumor tissue available for FISH testing [Wolff, 2007] in central laboratory
* Women and men with potential to have children must be willing to practice acceptable methods of birth control during the study
* Washout period from the prior last therapy as follows; Chemotherapy (except for agents below) 4 weeks (IV) Chemotherapy (except for agents below) 2 weeks (P.O) Trastuzumab, Bevacizumab 4 weeks Mitomycin-C, nitrosourea 6 weeks Radiotherapy, Immunotherapy, Biologic therapy and Surgery (except for minor surgical procedure) 2 weeks
* Willing to complete all screening assessments as outlined in the protocol
* Adequate organ function as defined in Table 2
* Gastrectomy status depending on the result in the Pilot Part
* Life expectancy of at least 12 weeks from the first dose of study treatment

Table 2 Baseline Laboratory Values

SYSTEM LABORATORY (VALUES)

Hematologic:

ANC (absolute neutrophil count)

Hemoglobin:

Platelets (≥ 2.0 × 10^9/L) (≥ 9 g/dL) (≥ 100 × 10^9/L) Hepatic Albumin Serum bilirubin AST and ALT (≥ 2.5 g/dL) (≤ 1.25 x ULN) (≤ 2.5 × ULN without liver metastases) (≤ 5 × ULN if documented liver metastases) Renal Serum Creatinine

Calculate Creatinine Clearance (see Section 11.3) (≤ 2.0 mg/dL)

- OR - (≥30 mL/min)

Exclusion criteria:

Subjects meeting any of the following criteria must not be enrolled in the study:

* Pregnant or lactating female at anytime during the study
* Planned concurrent anti-cancer therapy (chemotherapy, radiotherapy, immunotherapy, biologic therapy, hormonal therapy) while taking investigational treatment
* Unresolved or unstable, serious toxicity from prior cancer treatment (any toxicities greater than grade 2)
* Peripheral neuropathy of Grade 2 or greater
* Malabsorption syndrome, disease significantly affecting gastrointestinal function. Subjects with ulcerative colitis and Crohn's disease are also excluded
* History of other malignancy. However, subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma, are eligible
* Concurrent disease or condition that would make the subject inappropriate for study participation or any serious medical disorder that would interfere with the subject's safety
* Life threatening infection
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent
* Known history of uncontrolled or symptomatic angina, arrhythmias, or congestive heart failure
* Known history or clinical evidence of central nervous system (CNS) metastasis
* Concurrent treatment with prohibited medications, including herbal remedies and Chinese traditional medicines
* Concurrent treatment with an investigational agent within 28 days prior to the administration of paclitaxel and/or lapatinib
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to paclitaxel, including polyethoxylated castor oil, alcohol, or lapatinib or their excipients
* Anamnesis or diagnosis of pulmonary disorder, such as interstitial pneumonia, pulmonary fibrosis or serious hypoxia
* Gastrectomy surgery if Pilot Part of the study determines that partial gastrectomy (pylorus spared) or total/partial gastrectomy (pylorus removed) has a significant negative impact upon lapatinib PK and safety profile
* Known history of use of any EGFR agent (except Trastuzumab)
* Prior gastric cancer treatment which included a taxane.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2007-07; Primary Completion 2012-01 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- China (3):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Shanghai
- GSK Investigational Site, Tokyo, Japan
- South Korea (3):
  - GSK Investigational Site, Hwasun
  - GSK Investigational Site, Seongnam-si Gyeonggi-do
  - GSK Investigational Site, Seoul
- Taiwan (6):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Niaosong Township, Kaohsiung
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Tainan County
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Tau-Yuan County

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of a Pilot part and a Randomized part. The Pilot part and the Randomized part had two separate participant (par.) populations. The study period of the Randomized part was from 31 March 2008 to 5 January 2012 (cut-off date for efficacy). Follow-up was conducted until 30 October 2012 (cut-off date for safety analysis).
Pre-assignment Details: In the Pilot part, par. were enrolled in this study based on their gastrectomy status: non-gastrectomy (intact stomach), partial gastrectomy (gastrectomy with pylorus preserved), and gastrectomy (pylorus removed). However, no par. with partial gastrectomy were enrolled. In the Randomized part, par. were randomized to two treatment arms.
Groups:
- Lapatinib Plus Paclitaxel in Non-gastrectomy Participants: Participants with non-gastrectomy (intact stomach) received 1500 milligrams (mg) of oral lapatinib once daily throughout the study duration (lapatinib was not administered on Day 1 of the first cycle). Participants received a paclitaxel 1-hour intravenous infusion weekly for 3 weeks of a 4-week cycle at 80 mg per square meters (m^2).
- Lapatinib Plus Paclitaxel in Partial Gastrectomy Participants: Participants with partial gastrectomy (which includes preservation of the pylorus) received 1500 mg of oral lapatinib once daily throughout the study duration (lapatinib was not administered on Day 1 of the first cycle). Participants received a paclitaxel 1-hour intravenous infusion weekly for 3 weeks of a 4-week cycle at 80 mg/m^2. Partial gastrectomy (pylorus preserved) is very rare population in Japan. As a result, no such participants were recruited into this cohort.
- Lapatinib Plus Paclitaxel in Gastrectomy Participants: Participants with gastrectomy (pylorus removed) received 1500 mg of oral lapatinib once daily throughout the study duration (lapatinib was not administered on Day 1 of the first cycle). Participants received a paclitaxel 1-hour intravenous infusion weekly for 3 weeks of a 4-week cycle at 80 mg/m^2.
- Lapatinib Plus Paclitaxel: Participants received 1500 mg of oral lapatinib once daily throughout the study duration. Participants received a paclitaxel 1-hour intravenous infusion weekly for 3 weeks of a 4-week cycle at 80 mg/m^2 (on Days 1, 8, and 15 of each cycle).
- Paclitaxel Alone: Participants received a paclitaxel 1-hour intravenous infusion weekly for 3 weeks of a 4-week cycle at 80 mg/m^2 (on Days 1, 8, and 15 of each cycle).
Period: Pilot Part
Arm/Group | Lapatinib Plus Paclitaxel in Non-gastrectomy Participants | Lapatinib Plus Paclitaxel in Partial Gastrectomy Participants | Lapatinib Plus Paclitaxel in Gastrectomy Participants | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Started | 6 | 0 | 6 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 0 | 6 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 5 | 0 | 0
Not completed — Disease Progression | 2 | 0 | 1 | 0 | 0
Period: Randomized Part
Arm/Group | Lapatinib Plus Paclitaxel in Non-gastrectomy Participants | Lapatinib Plus Paclitaxel in Partial Gastrectomy Participants | Lapatinib Plus Paclitaxel in Gastrectomy Participants | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Started | 0 | 0 | 0 | 132 | 129
Completed | 0 | 0 | 0 | 112 | 115
Not Completed | 0 | 0 | 0 | 20 | 14
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0
Not completed — Sponsor Terminated Study | 0 | 0 | 0 | 19 | 13

BASELINE CHARACTERISTICS:
Groups:
- Lapatinib Plus Paclitaxel in Non-gastrectomy Participants: In the Pilot part, participants with non-gastrectomy (intact stomach) received 1500 milligrams (mg) of oral lapatinib once daily throughout the study duration (lapatinib was not administered on Day 1 of the first cycle). Participants received a paclitaxel 1-hour intravenous infusion weekly for 3 weeks of a 4-week cycle at 80 mg per square meters (m^2).
- Lapatinib Plus Paclitaxel in Gastrectomy Participants: In the Pilot part, participants with gastrectomy (pylorus removed) received 1500 mg of oral lapatinib once daily throughout the study duration (lapatinib was not administered on Day 1 of the first cycle). Participants received a paclitaxel 1-hour intravenous infusion weekly for 3 weeks of a 4-week cycle at 80 mg/m^2.
- Lapatinib Plus Paclitaxel in Randomized Part: Participants received 1500 mg of oral lapatinib once daily throughout the study duration. Participants received a paclitaxel 1-hour intravenous infusion weekly for 3 weeks of a 4-week cycle at 80 mg/m^2 (on Days 1, 8, and 15 of each cycle).
- Paclitaxel Alone in Randomized Part: Participants received a paclitaxel 1-hour intravenous infusion weekly for 3 weeks of a 4-week cycle at 80 mg/m^2 (on Days 1, 8, and 15 of each cycle).
- Total: Total of all reporting groups
Arm/Group | Lapatinib Plus Paclitaxel in Non-gastrectomy Participants | Lapatinib Plus Paclitaxel in Gastrectomy Participants | Lapatinib Plus Paclitaxel in Randomized Part | Paclitaxel Alone in Randomized Part | Total
Number analyzed (Participants) | 6 | 6 | 132 | 129 | 273
Age Continuous [Mean (Standard Deviation); unit: Years] | 57.5 (11.31) | 57.2 (10.98) | 60.8 (9.45) | 60.4 (10.96) | 60.5 (10.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 31 | 23 | 55
  Male | 5 | 6 | 101 | 106 | 218
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Japanese Heritage | 6 | 6 | 52 | 48 | 112
  Asian - East Asian Heritage | 0 | 0 | 73 | 75 | 148
  Asian - South East Asian Heritage | 0 | 0 | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) in the Pilot Part of the Study
Description: DLTs consisted of only drug-related toxicities (neurologic and non-neurologic DLTs). A neurologic DLT was defined as grade 3/4 clinically significant peripheral motor and/or sensitive neuropathy. Non-neurologic DLTs mainly included the following: grade 3/4 clinically significant non-hematological toxicity (except nausea), grade 4 neutropenia lasting >=7 days, thrombocytopenia (<=25000 cells per cubic millimeter), inability to begin next treatment within 2 weeks of scheduled dosing due to unresolved toxicity, treatment delay (due to toxicity) of >5 days, for Days 8 or 15 of weekly paclitaxel.
Time Frame: 28 days
Population: Safety Population (Pilot part): all participants who received at least one dose of investigational product in the Pilot part of the study
Measure: Number; unit: Participants
Arm/Group | Lapatinib Plus Paclitaxel in Non-gastrectomy Participants | Lapatinib Plus Paclitaxel in Gastrectomy Participants
Number analyzed (Participants) | 6 | 6
Participants | 2 | 1

2. Primary Outcome: Overall Survival (OS) in the Randomized Part of the Study
Description: OS was defined as the time from randomization until death due to any cause. For participants who did not die, time to death was censored at the time of last contact. For censored participants, time to death was defined as the time from randomization to the time of last contact.
Time Frame: From randomization until death due to any cause (up to 42.58 months)
Population: Intent-to-Treat Population: all participants who were randomized to study treatment, regardless of whether they actually received study medication
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 132 | 129
months | 11.0 [9.5 to 14.5] | 8.9 [7.4 to 11.1]
Statistical Analysis 1: Comparison: Lapatinib Plus Paclitaxel vs Paclitaxel Alone; Test type: Superiority or Other; p = 0.2088, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.64 to 1.11]

3. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Lapatinib in the Pilot Part of the Study
Description: Pharmacokinetic (PK) samples were collected at pre-dose and at 0.5, 1.0, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post dose on Days 8 and 14.
Time Frame: Days 8 and 14
Population: PK Parameter Population: all participants for whom the PK parameter could be estimated
Measure: Geometric Mean (95% Confidence Interval); unit: nanograms per milliliter (ng/mL)
Arm/Group | Lapatinib Plus Paclitaxel in Non-gastrectomy Participants | Lapatinib Plus Paclitaxel in Gastrectomy Participants
Number analyzed (Participants) | 6 | 6
nanograms per milliliter (ng/mL)
  Day 8 | 5435.525 [3932.949 to 7512.158] | 3129.561 [2429.401 to 4031.507]
  Day 14 | 3930.780 [3239.218 to 4769.988] | 2062.557 [1301.258 to 3269.251]

4. Secondary Outcome: Time to Cmax (Tmax) of Lapatinib in the Pilot Part of the Study
Description: PK samples were collected at pre-dose and at 0.5, 1.0, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post dose on Days 8 and 14.
Time Frame: Days 8 and 14
Population: PK Parameter Population
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | Lapatinib Plus Paclitaxel in Non-gastrectomy Participants | Lapatinib Plus Paclitaxel in Gastrectomy Participants
Number analyzed (Participants) | 6 | 6
hours (hr)
  Day 8 | 4.083 [2.98 to 8.00] | 3.500 [2.97 to 6.05]
  Day 14 | 7.992 [3.10 to 11.97] | 4.000 [3.03 to 4.08]

5. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to 24 Hours (AUC[0-24]) of Lapatinib in the Pilot Part of the Study
Description: PK samples were collected at pre-dose and at 0.5, 1.0, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post dose on Days 8 and 14. AUC is defined as the area under the lapatinib concentration-time curve as a measure of drug exposure. AUC(0-24) is area under the plasma concentration-time curve from time 0 to 24 hours after oral adminisation.
Time Frame: Days 8 and 14
Population: PK Parameter Population
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ng/mL
Arm/Group | Lapatinib Plus Paclitaxel in Non-gastrectomy Participants | Lapatinib Plus Paclitaxel in Gastrectomy Participants
Number analyzed (Participants) | 6 | 6
hr*ng/mL
  Day 8 | 86584.045 [71317.921 to 105117.994] | 37332.880 [27185.084 to 51268.700]
  Day 14 | 68177.402 [54550.364 to 85208.564] | 30565.248 [18109.123 to 51589.156]

6. Secondary Outcome: Cmax of Paclitaxel in the Pilot Part of the Study
Description: PK samples were collected just before the start of infusion and 0.5, 1.0 (immediately before terminating the infusion), 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post dose on Days 1 and 8.
Time Frame: Days 1 and 8
Population: PK Parameter Population
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Lapatinib Plus Paclitaxel in Non-gastrectomy Participants | Lapatinib Plus Paclitaxel in Gastrectomy Participants
Number analyzed (Participants) | 6 | 6
ng/mL
  Day 1 | 4121.513 [3524.391 to 4819.803] | 2731.104 [2275.497 to 3277.934]
  Day 8 | 4610.176 [3896.911 to 5453.992] | 2949.770 [2695.770 to 3227.702]

7. Secondary Outcome: Tmax of Paclitaxel in the Pilot Part of the Study
Description: as for outcome 6
Time Frame: Days 1 and 8
Population: PK Parameter Population
Measure: Median (Full Range); unit: hr
Arm/Group | Lapatinib Plus Paclitaxel in Non-gastrectomy Participants | Lapatinib Plus Paclitaxel in Gastrectomy Participants
Number analyzed (Participants) | 6 | 6
hr
  Day 1 | 1.042 [1.00 to 1.42] | 1.075 [0.98 to 1.25]
  Day 8 | 1.050 [1.00 to 1.18] | 1.025 [1.00 to 1.07]

8. Secondary Outcome: AUC(0-24) of Paclitaxel in the Pilot Part of the Study
Description: PK samples were collected just before the start of infusion and 0.5, 1.0 (immediately before terminating the infusion), 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post dose on Days 1 and 8. AUC is defined as the area under the paclitaxel concentration-time curve as a measure of drug exposure. AUC(0-24) is area under the plasma concentration-time curve from the start of infusion (time 0) to 24 hours after the start of the infusion.
Time Frame: Days 1 and 8
Population: PK Parameter Population
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ng/mL
Arm/Group | Lapatinib Plus Paclitaxel in Non-gastrectomy Participants | Lapatinib Plus Paclitaxel in Gastrectomy Participants
Number analyzed (Participants) | 6 | 6
hr*ng/mL
  Day 1 | 5771.847 [4726.425 to 7048.502] | 3968.654 [3531.979 to 4459.317]
  Day 8 | 7492.825 [6182.574 to 9080.754] | 4992.934 [4432.158 to 5624.660]

9. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUC[0-inf]) of Paclitaxel in the Pilot Part of the Study
Description: PK samples were collected just before the start of infusion and 0.5, 1.0 (immediately before terminating the infusion), 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post dose on Days 1 and 8. AUC is defined as the area under the paclitaxel concentration-time curve as a measure of drug exposure. AUC(0-inf) is area under the plasma concentration-time curve from the start of infusion (time 0) extrapolated to infinity.
Time Frame: Days 1 and 8
Population: PK Parameter Population
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ng/mL
Arm/Group | Lapatinib Plus Paclitaxel in Non-gastrectomy Participants | Lapatinib Plus Paclitaxel in Gastrectomy Participants
Number analyzed (Participants) | 6 | 6
hr*ng/mL
  Day 1 | 6262.157 [5042.138 to 7777.378] | 4058.648 [3952.209 to 5143.429]
  Day 8 | 8340.326 [6835.815 to 10175.970] | 6020.878 [4347.656 to 8338.049]

10. Secondary Outcome: Half-life of Paclitaxel in the Pilot Part of the Study
Description: PK samples were collected just before the start of infusion and 0.5, 1.0 (immediately before terminating the infusion), 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post dose on Days 1 and 8. Half-life is defined as the time required for the amount of the drug in the plasma to decrease by half.
Time Frame: Days 1 and 8
Population: PK Parameter Population
Measure: Geometric Mean (95% Confidence Interval); unit: hr
Arm/Group | Lapatinib Plus Paclitaxel in Non-gastrectomy Participants | Lapatinib Plus Paclitaxel in Gastrectomy Participants
Number analyzed (Participants) | 6 | 6
hr
  Day 1 | 10.128 [8.886 to 11.543] | 13.053 [10.266 to 16.597]
  Day 8 | 10.342 [8.460 to 12.642] | 13.978 [7.748 to 25.219]

11. Secondary Outcome: Clearance of Paclitaxel in the Pilot Part of the Study
Description: PK samples were collected just before the start of infusion and 0.5, 1.0 (immediately before terminating the infusion), 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post dose on Days 1 and 8. Clearance is defined as the clearance of drug from plasma, which is defined as the volume of plasma from which drug is removed per unit time.
Time Frame: Days 1 and 8
Population: PK Parameter Population
Measure: Geometric Mean (95% Confidence Interval); unit: liters per hour per square meter
Arm/Group | Lapatinib Plus Paclitaxel in Non-gastrectomy Participants | Lapatinib Plus Paclitaxel in Gastrectomy Participants
Number analyzed (Participants) | 6 | 6
liters per hour per square meter
  Day 1 | 12.775 [10.286 to 15.866] | 17.744 [15.554 to 20.242]
  Day 8 | 9.592 [7.862 to 11.703] | 13.287 [9.595 to 18.401]

12. Secondary Outcome: Distribution Volume at Steady State (Vss) of Paclitaxel in the Pilot Part of the Study
Description: PK samples were collected just before the start of infusion and 0.5, 1.0 (immediately before terminating the infusion), 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post dose on Days 1 and 8. Vss is the volume of distribution at steady state of paclitaxel.
Time Frame: Days 1 and 8
Population: PK Parameter Population
Measure: Geometric Mean (95% Confidence Interval); unit: liters per square meter
Arm/Group | Lapatinib Plus Paclitaxel in Non-gastrectomy Participants | Lapatinib Plus Paclitaxel in Gastrectomy Participants
Number analyzed (Participants) | 6 | 6
liters per square meter
  Day 1 | 76.011 [67.170 to 86.015] | 141.196 [110.329 to 180.698]
  Day 8 | 71.223 [55.644 to 91.163] | 126.121 [79.776 to 199.391]

13. Secondary Outcome: Progression-free Survival (PFS) in the Randomized Part of the Study
Description: PFS was defined as the time from randomization until the earliest date of disease progression (PD) or death due to any cause. Per Response Evaluation Criteria in Solid Tumors (RECIST), version 1.0, PD is defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started, or the appearance of one or more new lesions.
Time Frame: From randomization until disease progression or death due to any cause (up to 42.35 months)
Population: ITT Population. For participants whose disease did not progress or who did not die, PFS was censored at the time of the last independently assessed radiological scan preceding the initiation of any alternate anti-cancer therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 132 | 129
months | 5.4 [3.9 to 5.7] | 4.4 [3.7 to 5.6]

14. Secondary Outcome: Time to Progression in the Randomized Part of the Study
Description: Time to progression was defined as the time from randomization until the earliest date of disease progression or death due to disease. Per RECIST, version 1.0, PD is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started, or the appearance of one or more new lesions.
Time Frame: From randomization until disease progression or death due to disease (up to 42.35 months )
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 132 | 129
months | 5.5 [3.9 to 5.8] | 4.4 [3.7 to 5.6]

15. Secondary Outcome: Percentage of Participants With Overall Response in the Randomized Part of the Study
Description: Overall response was defined as the percentage of participants achieving either complete response (CR) or partial response (PR). Per RECIST, version 1.0, CR was defined as the disappearance of all target lesions, and PR was defined as a greater than 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.
Time Frame: From randomization up to 5.62 months
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 132 | 129
Percentage of participants | 27 | 9

16. Secondary Outcome: Number of Participants With the Indicated Time to Response in the Randomized Part of the Study
Description: Time to response was defined as the time from randomization to CR (the disappearance of all target lesions) or PR (a greater than 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD). For participants who did not achieve a CR or PR, time to response was censored at the last assessment prior to other cancer therapies. For censored participants, time to response was defined as the time from randomization to the time of the last assessment prior to the administation of other cancer therapies.
Time Frame: up to 5.62 months
Population: ITT Population. Only those participants achieving a CR or PR were assessed.
Measure: Number; unit: Participants
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 35 | 11
Participants
  Weeks 1-8 | 13 | 5
  Weeks >8 - 16 | 20 | 3
  Weeks >16 - 24 | 1 | 3
  Weeks >24 - 32 | 1 | 0

17. Secondary Outcome: Duration of Response in the Randomized Part of the Study
Description: Duration of response was defined as the time from the first documented evidence of CR (the disappearance of all target lesions) or PR (a greater than 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD) until the first documented sign of disease progression (at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started, or the appearance of one or more new lesions) or death due to any cause, if sooner.
Time Frame: up to 18.27 months
Population: ITT Population. Only those participants achieving a CR or PR were assessed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 35 | 11
months | 7.4 [5.0 to 11.0] | 5.1 [3.7 to 11.2]

18. Secondary Outcome: Number of Participants With the Indicated Grade 3 and Grade 4 Adverse Events (AEs) for Which All Grades of the AE Were Reported in >=10% of Participants, Regardless of Causality in the Randomized Part of the Study
Description: The Common Terminology Criteria for Advere Events (CTCAE) is a descriptive terminology that can be used for AE reporting. Grade (G) refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade (G) refers to the severity of the AE: G 1, mild AE; G 2, moderate AE; G 3, severe AE; G 4, life-threatening/disabling AE; G 5, death related to the AE.
Time Frame: From the first dose of investigational product to 30 days after the last dose (up to 110.3 weeks in the Randomized part)
Population: Safety Population: all participants who were randomized and took at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 131 | 129
participants
  Diarrhoea, Grade 3 | 23 | 3
  Diarrhoea, Grade 4 | 1 | 0
  Nausea, Grade 3 | 5 | 3
  Nausea, Grade 4 | 0 | 0
  Vomiting, Grade 3 | 4 | 4
  Vomiting, Grade 4 | 0 | 0
  Stomatitis, Grade 3 | 2 | 1
  Stomatitis, Grade 4 | 0 | 0
  Constipation, Grade 3 | 0 | 1
  Constipation, Grade 4 | 0 | 0
  Abdominal pain, Grade 3 | 0 | 0
  Abdominal pain, Grade 4 | 0 | 0
  Neutropenia, Grade 3 | 41 | 33
  Neutropenia, Grade 4 | 34 | 6
  Leukopenia, Grade 3 | 32 | 12
  Leukopenia, Grade 4 | 7 | 1
  Anaemia, Grade 3 | 10 | 8
  Anaemia, Grade 4 | 4 | 1
  Lymphopenia, Grade 3 | 4 | 2
  Lymphopenia, Grade 4 | 1 | 1
  Alopecia, Grade 3 | 0 | 0
  Alopecia, Grade 4 | 0 | 0
  Rash, Grade 3 | 3 | 0
  Rash, Grade 4 | 0 | 0
  Pruritus, Grade 3 | 0 | 0
  Pruritus, Grade 4 | 0 | 0
  Fatigue, Grade 3 | 6 | 1
  Fatigue, Grade 4 | 0 | 0
  Pyrexia, Grade 3 | 1 | 1
  Pyrexia, Grade 4 | 0 | 0
  Asthenia, Grade 3 | 1 | 0
  Asthenia, Grade 4 | 0 | 0
  Weight decreased, Grade 3 | 2 | 0
  Weight decreased, Grade 4 | 0 | 0
  White blood cell count decreased, Grade 3 | 18 | 6
  White blood cell count decreased, Grade 4 | 1 | 1
  Neutrophil count decreased, Grade 3 | 11 | 4
  Neutrophil count decreased, Grade 4 | 5 | 2
  Haemoglobin decreased, Grade 3 | 9 | 5
  Haemoglobin decreased, Grade (G) 4 | 1 | 0
  Aspartate aminotransferase increased, G 3 | 1 | 1
  Aspartate aminotransferase increased, G 4 | 1 | 0
  Alanine aminotransferase increased, G 3 | 2 | 2
  Alanine aminotransferase increased, G 4 | 1 | 0
  Peripheral sensory neuropathy, G 3 | 1 | 0
  Peripheral sensory neuropathy, G 4 | 0 | 0
  Neuropathy peripheral, Grade 3 | 2 | 1
  Neuropathy peripheral, Grade 4 | 0 | 0
  Decreased appetite, Grade 3 | 11 | 9
  Decreased appetite, Grade 4 | 1 | 0
  Myalgia, Grade 3 | 0 | 0
  Myalgia, Grade 4 | 0 | 0
  Arthralgia, Grade 3 | 2 | 0
  Arthralgia, Grade 4 | 0 | 0
  Back pain, Grade 3 | 0 | 0
  Back pain, Grade 4 | 0 | 0

19. Secondary Outcome: Change From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life (QOL) Questionnaire (EORTC QLQ-C30) Global Health Status (GHS)/QOL Score at the End of Therapy in the Randomized Part of the Study
Description: The EORTC QLQ-C30 is a 30-item, self-reporting questionnaire assessing 15 domains (5 functional scales [physical/role/emotional/cognitive/social]; 9 symptom scales [fatigue/nausea and vomiting/pain/dyspnea/insomnia/appetite loss/constipation/diarrhea/financial difficulties]; GHS/QOL scale). Participants assessed most statements on a 4-point scale (1, not at all; 4, very much); two questions used a 7-item scale (1, poor; 7, excellent). Scores were averaged and transformed to a 0-100 scale. A high score indicates both a high/healthy level of functioning and a high level of symptoms/problems.
Time Frame: Baseline and end of therapy (up to 42.58 months)
Population: ITT Population. Only those participants who contributed data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 90 | 70
scores on a scale | -12.41 (25.578) | -11.55 (28.562)

20. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Physical Functioning Score at the End of Therapy in the Randomized Part of the Study
Description: as for outcome 19
Time Frame: Baseline and end of therapy (up to 42.58 months)
Population: ITT Population. Only those participants who contributed data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 90 | 71
scores on a scale | -13.48 (18.776) | -13.99 (21.087)

21. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Role Functioning Score at the End of Therapy in the Randomized Part of the Study
Description: as for outcome 19
Time Frame: Baseline and end of therapy (up to 42.58 months)
Population: ITT Population. Only those participants who contributed data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 90 | 71
scores on a scale | -17.41 (24.468) | -18.31 (27.625)

22. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Emotional Functioning Score at the End of Therapy in the Randomized Part of the Study
Description: as for outcome 19
Time Frame: Baseline and end of therapy (up to 42.58 months)
Population: ITT Population. Only those participants who contributed data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 90 | 70
scores on a scale | -10.65 (19.594) | -10.12 (22.066)

23. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Cognitive Functioning Score at the End of Therapy in the Randomized Part of the Study
Description: as for outcome 19
Time Frame: Baseline and end of therapy (up to 42.58 months)
Population: ITT Population. Only those participants who contributed data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 90 | 70
scores on a scale | -10.19 (16.133) | -12.14 (20.446)

24. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Social Functioning Score at the End of Therapy in the Randomized Part of the Study
Description: as for outcome 19
Time Frame: Baseline and end of therapy (up to 42.58 months)
Population: ITT Population. Only those participants who contributed data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 90 | 70
scores on a scale | -10.74 (26.122) | -13.33 (22.089)

25. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Fatigue Symptom Score at the End of Therapy in the Randomized Part of the Study
Description: as for outcome 19
Time Frame: Baseline and end of therapy (up to 42.58 months)
Population: ITT Population. Only those participants who contributed data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 90 | 71
scores on a scale | 11.98 (21.084) | 14.79 (23.885)

26. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Nausea and Vomiting Symptom Score at the End of Therapy in the Randomized Part of the Study
Description: as for outcome 19
Time Frame: Baseline and end of therapy (up to 42.58 months)
Population: ITT Population. Only those participants who contributed data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 90 | 71
scores on a scale | 4.26 (17.411) | 7.28 (19.666)

27. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Pain Symptom Score at the End of Therapy in the Randomized Part of the Study
Description: as for outcome 19
Time Frame: Baseline and end of therapy (up to 42.58 months)
Population: ITT Population. Only those participants who contributed data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 90 | 71
scores on a scale | 7.41 (27.038) | 12.68 (29.743)

28. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Dyspnea Symptom Score at the End of Therapy in the Randomized Part of the Study
Description: as for outcome 19
Time Frame: Baseline and end of therapy (up to 42.58 months)
Population: ITT Population. Only those participants who contributed data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 90 | 71
scores on a scale | 12.22 (22.037) | 15.02 (23.764)

29. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Insomnia Symptom Score at the End of Therapy in the Randomized Part of the Study
Description: as for outcome 19
Time Frame: Baseline and end of therapy (up to 42.58 months)
Population: ITT Population. Only those participants who contributed data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 90 | 71
scores on a scale | 5.56 (28.813) | 10.80 (27.473)

30. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Appetite Loss Symptom Score at the End of Therapy in the Randomized Part of the Study
Description: as for outcome 19
Time Frame: Baseline and end of therapy (up to 42.58 months)
Population: ITT Population. Only those participants who contributed data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 90 | 71
scores on a scale | 12.59 (28.521) | 7.04 (28.683)

31. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Constipation Symptom Score at the End of Therapy in the Randomized Part of the Study
Description: as for outcome 19
Time Frame: Baseline and end of therapy (up to 42.58 months)
Population: ITT Population. Only those participants who contributed data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 90 | 71
scores on a scale | 5.93 (27.176) | 2.35 (26.621)

32. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Diarrhea Symptom Score at the End of Therapy in the Randomized Part of the Study
Description: as for outcome 19
Time Frame: Baseline and end of therapy (up to 42.58 months)
Population: ITT Population. Only those participants who contributed data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 90 | 70
scores on a scale | 10.00 (31.385) | 4.29 (24.025)

33. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Financial Difficulties Symptom Score at the End of Therapy in the Randomized Part of the Study
Description: as for outcome 19
Time Frame: Baseline and end of therapy (up to 42.58 months)
Population: ITT Population. Only those participants who contributed data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 90 | 70
scores on a scale | 7.04 (28.042) | 0.95 (27.200)

34. Secondary Outcome: Change From Baseline in the EORTC QLQ-STO22 Dysphagia Scale Score at the End of Therapy in the Randomized Part of the Study
Description: The EORTC QLQ-STO22 is a 22-item, self-reporting instrument consisting of 5 scales and 4 single items to assess health-related quality of life (HRQOL) issues related to dysphagia, eating restrictions, reflux, and abdominal pain, as well as specific symptoms that may occur during chemotherapy or radiation treatment. Scores are averaged and transformed to a 0-100 scale. For the symptom scales and items, a high score is equivalent to worse or more symptoms. In the functional scales, however, a high score is equivalent to better function.
Time Frame: Baseline and end of therapy (up to 42.58 months)
Population: ITT Population. Only those participants who contributed data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 90 | 71
scores on a scale | 10.37 (21.382) | 5.16 (14.887)

35. Secondary Outcome: Change From Baseline in the EORTC QLQ-STO22 Pain Scale Score at the End of Therapy in the Randomized Part of the Study
Description: as for outcome 34
Time Frame: Baseline and end of therapy (up to 42.58 months)
Population: ITT Population. Only those participants who contributed data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 90 | 71
scores on a scale | 5.46 (16.151) | 3.40 (14.542)

36. Secondary Outcome: Change From Baseline in the EORTC QLQ-STO22 Reflux Symptoms Scale Score at the End of Therapy in the Randomized Part of the Study
Description: as for outcome 34
Time Frame: Baseline and end of therapy (up to 42.58 months)
Population: ITT Population. Only those participants who contributed data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 90 | 71
scores on a scale | 3.33 (14.177) | 2.66 (15.312)

37. Secondary Outcome: Change From Baseline in the EORTC QLQ-STO22 Eating Restrictions Scale Score at the End of Therapy in the Randomized Part of the Study
Description: as for outcome 34
Time Frame: Baseline and end of therapy (up to 42.58 months)
Population: ITT Population. Only those participants who contributed data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 90 | 71
scores on a scale | 8.33 (18.780) | 6.69 (18.720)

38. Secondary Outcome: Change From Baseline in the EORTC QLQ-STO22 Anxiety Scale Score at the End of Therapy in the Randomized Part of the Study
Description: as for outcome 34
Time Frame: Baseline and end of therapy (up to 42.58 months)
Population: ITT Population. Only those participants who contributed data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 90 | 71
scores on a scale | 8.27 (24.624) | 2.97 (21.899)

39. Secondary Outcome: Change From Baseline in the EORTC QLQ-STO22 Dry Mouth Scale Score at the End of Therapy in the Randomized Part of the Study
Description: as for outcome 34
Time Frame: Baseline and end of therapy (up to 42.58 months)
Population: ITT Population. Only those participants who contributed data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 90 | 71
scores on a scale | 8.15 (27.053) | 2.35 (21.324)

40. Secondary Outcome: Change From Baseline in the EORTC QLQ-STO22 Taste Scale Score at the End of Therapy in the Randomized Part of the Study
Description: as for outcome 34
Time Frame: Baseline and end of therapy (up to 42.58 months)
Population: ITT Population. Only those participants who contributed data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 90 | 71
scores on a scale | 13.70 (28.659) | 3.29 (0)

41. Secondary Outcome: Change From Baseline in the EORTC QLQ-STO22 Body Image Scale Score at the End of Therapy in the Randomized Part of the Study
Description: as for outcome 34
Time Frame: Baseline and end of therapy (up to 42.58 months)
Population: ITT Population. Only those participants who contributed data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 90 | 71
scores on a scale | 15.99 (27.442) | 8.45 (32.229)

42. Secondary Outcome: Change From Baseline in the EORTC QLQ-STO22 Hair Loss Scale Score at the End of Therapy in the Randomized Part of the Study
Description: as for outcome 34
Time Frame: Baseline and end of therapy (up to 42.58 months)
Population: ITT Population. Only those participants who contributed data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 22 | 13
scores on a scale | 9.09 (31.171) | 7.69 (33.758)

43. Secondary Outcome: Number of Participants With the Indicated Epidermal Growth Factor Receptor (EGFR) Immunohistochemistry Intensity in the Randomized Part of the Study
Description: EGFR protein expression on the surface of cells in gastric cancer tissue samples was measured using a moncolonal antibody specific for the extracellular region of EGFR, and the degree of membrane staining was evaluated. 3+ indicates positive EGFR expression; <3+ indicates negative EGFR expression.
Time Frame: Pretreatment
Population: ITT Population. Only those participants for whom immunohistochemistry testing was conducted were analyzed.
Measure: Number; unit: participants
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 73 | 65
participants
  <3+ | 68 | 59
  3+ | 5 | 6

44. Secondary Outcome: Number of Participants With the Indicated Human Epidermal Growth Factor Receptor 2 (HER2) Immunohistochemistry Intensity in the Randomized Part of the Study
Description: HER2 protein expression on the surface of cells in gastric cancer tissue samples was measured using a monoclonal antibody specific for the extracellulr region of HER2, and the degree of membrane staining was evaulated. The immunohistochemistry test gives a score of 0 to 3+ and measures the amount of HER2 receptor protein on the surface of cells in a gastric cancer tissue sample. Score of 0 to 1+, "HER2 negative"; score of 2+, "borderline"; score of 3+, "HER2 positive."
Time Frame: Pretreatment
Population: ITT Population. Only those participants for whom immunohistochemistry testing was conducted were analyzed.
Measure: Number; unit: participants
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 100 | 92
participants
  0/1+ | 36 | 32
  2+ | 12 | 11
  3+ | 52 | 49

45. Secondary Outcome: Number of Participants With Mutations That May Correlate With Response and Toxicity to Lapatinib
Description: An inadequate number of tissue samples were obtained; thus, analysis could not be performed.
Time Frame: Pretreatment
Population: ITT Population
Arm/Group | Lapatinib Plus Paclitaxel | Paclitaxel Alone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the first dose of investigational product to 30 days after the last dose (up to 51.7 weeks in the Pilot part and up to 110.3 weeks in the Randomized part).
Description: SAEs and non-serious AEs were collected in members of the Safety Population in both the Pilot part and the Randomized part . For the Pilot part, MedDRA 12.1 was used; for the Randomized part, MedDRa 15.1 was used.
Arm/Group | Lapatinib Plus Paclitaxel in Non-gastrectomy Participants | Lapatinib Plus Paclitaxel in Gastrectomy Participants | Lapatinib Plus Paclitaxel in Randomized Part | Paclitaxel Alone in Randomized Part
Serious Adverse Events (participants affected / at risk) | 3/6 | 2/6 | 38/131 | 20/129
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 131/131 | 126/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib Plus Paclitaxel in Non-gastrectomy Participants (N=6) | Lapatinib Plus Paclitaxel in Gastrectomy Participants (N=6) | Lapatinib Plus Paclitaxel in Randomized Part (N=131) | Paclitaxel Alone in Randomized Part (N=129)
Pneumonia (Infections and infestations) | 0 | 1 | 2 | 4
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 3 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Beta haemolytic streptococcal infection (Infections and infestations) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 2 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 1
Infection (Infections and infestations) | 0 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Cholangitis suppurative (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 8 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 4 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib Plus Paclitaxel in Non-gastrectomy Participants (N=6) | Lapatinib Plus Paclitaxel in Gastrectomy Participants (N=6) | Lapatinib Plus Paclitaxel in Randomized Part (N=131) | Paclitaxel Alone in Randomized Part (N=129)
Neutropenia (Blood and lymphatic system disorders) | 6 | 5 | 85 | 64
Anaemia (Blood and lymphatic system disorders) | 5 | 1 | 45 | 27
Leukopenia (Blood and lymphatic system disorders) | 5 | 4 | 67 | 54
Lymphopenia (Blood and lymphatic system disorders) | 5 | 3 | 17 | 15
Monocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 1
Nausea (Gastrointestinal disorders) | 6 | 1 | 46 | 35
Diarrhoea (Gastrointestinal disorders) | 5 | 5 | 100 | 29
Stomatitis (Gastrointestinal disorders) | 3 | 2 | 41 | 18
Vomiting (Gastrointestinal disorders) | 3 | 1 | 38 | 23
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 6 | 3
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 8 | 7
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 1 | 5 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 15 | 26
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 17 | 8
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 10 | 8
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 9 | 2
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2 | 80 | 41
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 2 | 10 | 5
Hypoproteinaemia (Metabolism and nutrition disorders) | 2 | 1 | 3 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 9 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 3 | 5
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 6 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 3
Dysgeusia (Nervous system disorders) | 2 | 3 | 15 | 5
Headache (Nervous system disorders) | 2 | 1 | 9 | 4
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 13 | 7
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 19 | 20
Myoclonus (Nervous system disorders) | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 3 | 33 | 28
Somnolence (Nervous system disorders) | 1 | 2 | 3 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 12 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 4 | 88 | 73
Rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 64 | 19
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 12 | 4
Nail disorder (Skin and subcutaneous tissue disorders) | 2 | 0 | 15 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 23 | 11
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 10 | 3
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 4 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 4 | 2 | 36 | 16
Fatigue (General disorders) | 3 | 4 | 56 | 48
Chills (General disorders) | 1 | 0 | 0 | 3
Oedema (General disorders) | 1 | 1 | 5 | 3
Thirst (General disorders) | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 3 | 5
Oedema peripheral (General disorders) | 0 | 1 | 6 | 8
Asthenia (General disorders) | 0 | 0 | 20 | 8
Malaise (General disorders) | 0 | 0 | 8 | 4
Alanine aminotransferase increased (Investigations) | 3 | 4 | 16 | 11
Aspartate aminotransferase increased (Investigations) | 3 | 3 | 14 | 14
Blood alkaline phosphatase increased (Investigations) | 3 | 3 | 10 | 7
Blood albumin decreased (Investigations) | 2 | 0 | 6 | 2
Blood chloride decreased (Investigations) | 2 | 0 | 0 | 0
Blood urine present (Investigations) | 2 | 0 | 2 | 2
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 2 | 0
Blood amylase increased (Investigations) | 1 | 0 | 0 | 0
Blood calcium decreased (Investigations) | 1 | 0 | 3 | 2
Blood creatinine increased (Investigations) | 1 | 0 | 5 | 1
Blood potassium decreased (Investigations) | 1 | 1 | 7 | 0
Blood urea increased (Investigations) | 1 | 0 | 3 | 0
Glucose urine present (Investigations) | 1 | 1 | 2 | 3
Monocyte count decreased (Investigations) | 1 | 0 | 2 | 1
Platelet count increased (Investigations) | 1 | 1 | 2 | 0
Protein urine present (Investigations) | 1 | 0 | 1 | 1
Specific gravity urine decreased (Investigations) | 1 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 2 | 49 | 29
Haemoglobin decreased (Investigations) | 0 | 2 | 20 | 19
Blood bilirubin increased (Investigations) | 0 | 1 | 6 | 7
Blood chloride increased (Investigations) | 0 | 1 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 28 | 25
Neutrophil count decreased (Investigations) | 0 | 0 | 23 | 18
Biliary dilatation (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 7 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 3 | 8 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 21 | 22
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 16 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 14 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 11 | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 22 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 9 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 7 | 2
Infection (Infections and infestations) | 1 | 1 | 7 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 10 | 9
Paronychia (Infections and infestations) | 1 | 0 | 13 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 4 | 4
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Neutropenic infection (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 10 | 5
Insomnia (Psychiatric disorders) | 2 | 3 | 10 | 8
Proteinuria (Renal and urinary disorders) | 2 | 0 | 5 | 2
Dysuria (Renal and urinary disorders) | 1 | 0 | 2 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 0
Post gastric surgery syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.